CLINICAL TRIAL: NCT06294522
Title: Lecturer of Oral and Maxillofacial Surgery
Brief Title: Reconstruction of Nasal Floor for Three-dimensional Repair of Alveolar Cleft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, mona samy sheta, lecturer of oral and maxillofacial surgery department, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1984
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Alveolar Cleft
Keywords: alveolar cleft; nasal floor support; autogenous bone graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- reconstruction of alveolar cleft (Experimental): gingival mucoperiosteal flaps are designed along the cleft margins and elevated. These flaps are raised up and then are separated from the nasal mucosa the palatal mucoperiosteal flaps along the cleft margins are then elevated from the palate. After complete exposure of all the bony clefts, the nasal lining of the nostril floor is approximated and sutured, and the palatal flaps are then turned back and sutured to make a soft-tissue pocket. Grafting of the defect is accomplished with cortical bone only from the chin the cortical shelf is prepared to be two layers perpendicular to each other the first one is parallel to the nasal floor and second one is continuous with buccal cortex of alveolar ridge then cancellous bone will be packed under these shelves and be compressed into the cleft defects.
  Interventions: Procedure: reconstruction of alveolar cleft

INTERVENTIONS:
Procedure: reconstruction of alveolar cleft — after elevation of mucoperiosteal flap related to cleft side. suturing of nasal floor and palatal tissue. harvesting of autogenous graft and reconstruction of nasal floor and labial plate of cleft then suturing of flap labially without tension

SUMMARY:
reconstruction of alveolar cleft with autogenous bone after elevation of mucoperiosteal flap and suturing of nasal floor and palatal flap

DETAILED DESCRIPTION:
gingival mucoperiosteal flaps are designed along the cleft margins and elevated medial and lateral mucoperiosteal flaps are generated from the cleft and the gingival sulcus of the teeth. To obtain adequate mobility of the posterior flap, the flap must be extended to the first or the second molar and back-cut up to the buccal sulcus while taking care not to injure the alveolar bone covering the roots of the teeth. These flaps are raised up to and around the piriform aperture, and then are separated from the nasal mucosa the palatal mucoperiosteal flaps along the cleft margins are then elevated from the palate. After complete exposure of all the bony clefts, the nasal lining of the nostril floor is approximated and sutured, and the palatal flaps are then turned back and sutured to make a soft-tissue pocket. Grafting of the defect is accomplished with cortical bone only from the chin the cortical shelf is prepared to be two layers perpendicular to each other the first one is parallel to the nasal floor and second one is continuous with buccal cortex of alveolar ridge then cancellous bone will be packed under these shelves and be compressed into the cleft defect to maximize the number of osteo-competent cells and the osteoid material per unit graft volume. When packing bone particles, it is better to create the maxilla and alveolar ridges and elevate the depressed nostril by appropriately supporting the nasal base and aligning the symmetry. The rest can then be covered with gingival mucoperiosteal flaps through tension-free transposition

ELIGIBILITY:
Inclusion Criteria:

patients had alveolar cleft adequate and healthy soft tissue

-

Exclusion Criteria:

* age less than 9 very wide cleft scared soft tissue

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
recurrence of oronasal fistula | one month
  using valsalva test
volume of alveolar cleft after reconstruction | immediate and after 6 months
  using cone beam ct (cbct) to measure volumetric changes
density of bone | Six months
  using cbct with housenfield units D1 (>1250), D2(850-1250),D3(350-850),D4(150-350)

CONTACTS AND LOCATIONS:
Overall Officials: mona s sheta, Principal Investigator — Tanta University
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt